CLINICAL TRIAL: NCT02595203
Title: A Phase I, Two-part, Open-label, Non-randomised Study to Investigate the Mass Balance Recovery and Metabolic Profile of 14C Debio 1450 Following Single Oral and Intravenous Doses in Healthy Male Subjects
Brief Title: Mass Balance Recovery and Metabolic Profile of 14C Debio 1450 Following Single Oral and Intravenous Doses in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Debio 1450-105; 2015-002604-87 (EudraCT Number)
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A: Cohort 1 (Experimental): Participants receive a single intravenous (IV) dose of 240 mg/3.7 megabecquerel (MBq) of [14C-pos 1]-Debio 1450 BES solution.
  Interventions: Drug: [14C-pos 1]-Debio 1450 BES Solution
- Part A: Cohort 2 (Experimental): Participants receive a single oral dose of 240 mg/3.7 MBq of [14C-pos 1]-Debio 1450 BES solution.
  Interventions: Drug: [14C-pos 1]-Debio 1450 BES Solution
- Part B: Cohort 3 (Experimental): Participants receive a single oral dose of 240 mg Debio 1450/37 kilobecquerel (kBq) of [14C-pos 25]-Debio 1450 BES solution.
  Interventions: Drug: [14C-pos 25]-Debio 1450 BES Solution

INTERVENTIONS:
Drug: [14C-pos 1]-Debio 1450 BES Solution — A solution containing Debio 1450 bis ethanolamine salt (BES) radiolabelled with carbon-14 (14C) at position 1
  Arms: Part A: Cohort 1; Part A: Cohort 2
Drug: [14C-pos 25]-Debio 1450 BES Solution — A solution containing Debio 1450 BES radiolabelled with carbon-14 (14C) at position 25
  Arms: Part B: Cohort 3

SUMMARY:
The primary objectives of this study are:

* To determine the mass balance recovery (expired air, urine and faeces) and route and rate of elimination of 14C-Debio 1450.
* To determine the metabolic profile of 14C-Debio 1450 in whole blood, plasma, urine and faeces.
* To determine the pharmacokinetics of total radioactivity and of Debio 1450 (prodrug) and Debio 1452 (active moiety) in plasma and urine.

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification and contraception
* Is willing and able to remain confined in the study unit for the entire duration of each treatment period and comply with restrictions related to food, drink and medications
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* Has history or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Has signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding)
  3. the analysis of results

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery after a single dose of radiolabelled Debio 1450 measured through total radioactivity excreted in expired air, urine and faeces | 168 hours after dosing (Day 8)
Routes of metabolism and excretion after a single dose of radiolabelled Debio 1450 measured through total radioactivity concentrations in expired air, urine and fecaes | 168 hours after dosing (Day 8)
Whole blood and plasma partitioning of total radioactivity after a single dose of radiolabelled Debio 1450 through measurement of total radioactivity levels in blood | 168 hours after dosing (Day 8)
  Blood is collected within the 168 hours as follows:
  * IV infusion: Predose, 1, 1.85, 2.25, 2.5, 3, 4, 5, 8, 14, 18, 24, 36, 48, 60, 72, 96, 120, 144 and 168 hours after the infusion start time
  * Oral administration: Predose,15 and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120, 144 and 168 hours following the oral dose
Percentage of participants with clinically significant change from baseline in vital signs, electrocardiogram, and/or laboratory parameters | 168 hours after dosing (Day 8)

CONTACTS AND LOCATIONS:
Overall Officials: Annick Ménétrey, Study Director — Debiopharm International, S.A.
Locations (1):
- Covance Clinical Research Unit (CRU) Ltd., Leeds, United Kingdom